CLINICAL TRIAL: NCT04471766
Title: Evaluation of Locally Produced Cloth Face Mask on COVID-19 and Respiratory Illnesses Prevention at the Community Level - a Cluster-randomized Trial
Brief Title: Locally Produced Cloth Face Mask and COVID-19 Like Illness Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bandim Health Project (Other)
Collaborators: University of Southern Denmark (Other); Engineers without Borders, Denmark (https://iug.dk/en) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BHP MASK01
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-03

CONDITIONS: COVID-19; Respiratory Illness
Keywords: Face mask; COVID-19; Respiratory illness; Mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Certified cloth face mask plus preventive information (Experimental): Certified cloth face mask
  Interventions: Other: Certified cloth face mask plus preventive information; Behavioral: Preventive information
- Information on COVID-19 prevention (Active Comparator): Advice on how to prevent COVID-19 according to the government´ policy.
  Interventions: Behavioral: Preventive information

INTERVENTIONS:
Other: Certified cloth face mask plus preventive information — Provision of two face masks sewed locally following a certified model tested for FORCE in the laboratory per residents > 10 years old
  Arms: Certified cloth face mask plus preventive information
Behavioral: Preventive information — Advice on how to prevent COVID-19 according to the government´ policy

SUMMARY:
The number of cases of COVID-19 is still increasing and transmission of SARS-CoV-2 seems to occur mainly through person-to-person transmission through respiratory droplets, indirect contact with infected people and surfaces. The use of face masks is recommended as a public health measure, but in many settings only domestic cloth made masks are available to the majority of the people. However, masks can be of different quality and very little is known about the utility of cloth face masks at the community level.

In Bandim Health Project's Health and Demographic Surveillance System we will evaluate the effect of providing locally produced cloth face masks on severity of COVID-19 like illness and mortality in an urban population. The locally produced cloth mask is made according to a laboratory certified model and will be provided to the intervention group alongside information of how the risk of transmission can be reduced. The control group will receive information alone.

Follow-up will be implemented through telephone calls and post-epidemic home visits.

ELIGIBILITY:
Inclusion Criteria:

* Household resident
* Age: 10 years and older

Exclusion Criteria:

* Refusal to participate

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40000 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Reported COVID-like illness | Four months follow-up
  Self-reported main symptoms of COVID-19 (three or more - fever, cough, fatigue, shortness of breath, loss of smell / taste)
Consultation | Four months follow-up
  Consultation for COVID-19 like illness or/and reported positive test
Severe illness | Four months follow-up
  Self reported COVID-19 like illness plus hospitalization or death
Mortality | Four months follow-up
  Any death during the follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Bandim Health Project, Bissau, Bissau Codex, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nanque LM, Jensen AM, Diness A, Nielsen S, Cabral C, Cawthorne D, Martins JSD, Ca EJC, Jensen K, Martins CL, Rodrigues A, Fisker AB. Effect of distributing locally produced cloth facemasks on COVID-19-like illness and all-cause mortality-a cluster-randomised controlled trial in urban Guinea-Bissau. PLOS Glob Public Health. 2024 Feb 13;4(2):e0002901. doi: 10.1371/journal.pgph.0002901. eCollection 2024. PMID 38349910

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT04471766/SAP_000.pdf